CLINICAL TRIAL: NCT07130877
Title: EFFICACY AND SAFETY OF F100 PREPARED BY RECIPE METHOD FOR WEIGHT GAIN IN SEVERELY ACUTE MALNOURISHED CHILDREN
Brief Title: RECIPE BASED F100 INTERVENTION FOR NUTRITIONAL EFFICACY IN SAM (REFINE-SAM )
Acronym: REFINE-SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital and Institute of Child Health, Multan (Other Government)
Responsible Party: Principal Investigator, Dr. Saadia Khan, Principal Investigator, Children's Hospital and Institute of Child Health, Multan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1326-4619
Record Dates: First submitted 2025-08-07; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Severe Acute Malnutrition
Keywords: F100; Recipe-based formula; Therapeutic feeding
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WHO F-100 Formula (Active Comparator): WHO already made formula will be given after initial stabilization starting from 150 kcal per kg per day to a maximum of 220 kcal per kg per day at 4-hourly intervals, and intakes and vitals will be monitored.
  Interventions: Dietary Supplement: WHO F100
- WHO RECIPE MADE F100 (Experimental): Who recipe made F100 formula will be given after initial stabilization, starting from 150 kcal per kg per day to a maximum of 220 kcal per kg per day at 4-hourly intervals, and intakes and vitals will be monitored.
  Interventions: Dietary Supplement: WHO RECIPE BASED F100

INTERVENTIONS:
Dietary Supplement: WHO F100 — WHO F1OO
  Arms: WHO F-100 Formula
Dietary Supplement: WHO RECIPE BASED F100 — Recipe-made formula will be given after initial stabilization, starting from 150 kcal per kg per day to a maximum of 220 kcal per kg per day at 4-hourly intervals, and intakes and vitals will be monitored.
  Arms: WHO RECIPE MADE F100

SUMMARY:
This open-label randomized controlled trial evaluates the efficacy and safety of multiple formulations of the F-100 therapeutic feed during the rehabilitation phase among children aged 6-59 months with SAM, in comparison to standard WHO F-100. The primary outcome is daily weight gain (g/kg/day) over 10 days; secondary outcomes include MUAC improvement, gastrointestinal tolerance (vomiting/diarrhea), duration to recovery, and renal safety markers (serum urea, creatinine, serum sodium, urine-specific gravity).

DETAILED DESCRIPTION:
This open-label randomized controlled trial evaluates the efficacy and safety of multiple formulations of the F-100 therapeutic feed during the rehabilitation phase among children aged 6-59 months with SAM, in comparison to standard WHO F-100. The study includes four arms: the WHO commercial F-100 powder (control), recipe-based locally prepared F-100 (Arm A), diluted F-100 (Arm B), and an alternative locally prepared high-energy RUTF-like blend (Arm C). The primary outcome is daily weight gain (g/kg/day) over 10 days; secondary outcomes include MUAC improvement, gastrointestinal tolerance (vomiting/diarrhea), duration to recovery, and renal safety markers (serum urea, creatinine, serum sodium, urine-specific gravity).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-59 months
* Diagnosed with SAM
* Have completed stabilization and entering rehabilitation phase per WHO CMAM guidelines

Exclusion Criteria:

* Secondary malnutrition (e.g. tuberculosis, HIV)
* Chronic systemic diseases
* Congenital anomalies
* Terminal illness

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mean weight gain (g/kg/day) during rehabilitation | From randomization to after starting treatment 10 days
  Mean weight gain (g/kg/day) during 10 days of rehabilitation

SECONDARY OUTCOMES:
MUAC | From randomization to after starting treatment 10 days
  Improvement of F MUAC
Safety profile | From randomization to after starting treatment 10 days
  Incidence of treatment-related adverse events (nausea, vomiting, and fluid overload) assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Acceptability and Palatability by Hedonic scale scores for taste and acceptability of F-100 | day 1
  Palatability assessed using a 5-point Hedonic Scale adapted for pediatric populations. Scores collected on day 1
Change in serum albumin levels from baseline to day 10 | base line and day 10
  Serum albumin measured in g/dL using a standard automated biochemical analyzer. Change calculated as day 10 value minus baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad T Sultan, PhD, Study Chair — Bahuddin Zakariya University,Multan.
Locations (2):
- Pakistan (2):
  - Children's Hospital and Institute of child health Multan, Multan, Punjab Province
  - Tehsil Head Quater Sujah Abad, Multan Khurd, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Munirul Islam MM, Dafni M, et al. Efficacy of F-100, diluted F-100 (F100D), and infant formula as rehabilitation diet for infants aged < 6 months with severe acute malnutrition: a randomized clinical trial. Eur J Nutr. 2020 — https://pubmed.ncbi.nlm.nih.gov/36438193/